CLINICAL TRIAL: NCT06057545
Title: A Multi-center Interventional Study to Assess Pharmacokinetics, Effectiveness and Tolerability of Prolonged-release Tacrolimus After Paediatric Kidney Transplantation
Brief Title: Pharmacokinetics, Effectiveness and Tolerability of Prolonged-release Tacrolimus After Paediatric Kidney Transplantation
Acronym: Pro-Tac
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro-Tac
Record Dates: First submitted 2023-04-24; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Pediatric Kidney Disease
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, interventional, open-label, randomized, two-phase, two-sequence, single dose, crossover, phase III b
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Envarsus followed by Prograf (Experimental): 4 weeks treatment sequence 1 (Envarsus) followed by 4 weeks treatment sequence 2 (Prograf)
  Interventions: Drug: Envarsus®; Drug: Prograf
- Group B - Prograf followed by Envarsus (Experimental): 4 weeks treatment sequence 2 (Prograf) followed by 4 weeks treatment sequence 1 (Envarsus)
  Interventions: Drug: Envarsus®; Drug: Prograf

INTERVENTIONS:
Drug: Envarsus® — Treatment sequence: 4 weeks prolonged-release tacrolimus (Envarsus®) once daily
Drug: Prograf — Treatment sequence: 4 weeks intermediate-release tacrolimus (Prograf®) twice daily

SUMMARY:
Recently, a new prolonged-release tablet version of tacrolimus (Envarsus®) using the so-called MeltDose™ (US Patent No. 7,217,431) drug-delivery technology has been approved as immunosuppressive medication for patients after kidney and liver transplantation in adults but not yet in children. Studies in adults proved that Envarsus® provides the same therapeutic effectiveness as the conventional immediate-release tacrolimus formulation (Prograf®) with improved bioavailability, a more consistent pharmacokinetic profile and reduced peak to trough which might result in reduced tacrolimus dosing and subsequently reduced CNI related toxicity. Furthermore, the once daily formulation might result in improved drug adherence.

The aim of this study is to assess pharmacokinetic profiles of Envarsus® as well as effectiveness and tolerability of this drug in children and adolescents ≥ 8 and ≤ 18 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. caucasian paediatric kidney transplant recipients (single-organ recipients)
2. aged ≥ 8 years but ≤ 18 years who are under tacrolimus (Prograf®) therapy and who are able to swallow tablets with a minimum dose of 0.75 mg / day Envarsus®
3. not less than 6 months after transplantation
4. stable kidney function (delta eGFR < 10 ml/min/1.73 m2 (CKID formula) over the last 3 months)
5. women of childbearing potential and women without childbearing potential
6. patient/parents/legal guardian(s) must be capable of understanding purpose and risks of the study
7. signed informed consent obtained by patient and parents/legal guardians

Exclusion Criteria:

1. coefficient of variation of tacrolimus trough levels > 0.35 over the previous 6 months
2. pregnancy/breast feeding
3. instable kidney function
4. hypersensitivity to any of the components of the medications used
5. not eligible for any reason according to the investigator's valuation
6. known positive HIV-1 or HCV test
7. participation in another clinical trial (other investigational drugs or devices at the time of enrolment or within 30 days prior to enrolment)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Full tacrolimus AUC | 4 weeks
  full tacrolimus AUC calculated from Tac measures before administration of drug and 1.5, 2, 4, 6, 8, 12, 13.5, 14, 16, 20, 24 hours after administration of drug at the time point of 2 weeks (14±7 days) after end of build-up period for each patient under both treatments within two time periods with each a length of 4 weeks

SECONDARY OUTCOMES:
Pharmacodynamic analysis | 4 weeks
  Assessment of efficacy in terms of residual expression of NFAT regulated genes, expressed as % of expression at C0 (time point before drug administration set at 100%) at 1.5, 2, 4, 6, 8, 12, 13.5, 14, 16, 20, 24 hours after administration of drug at the time point of 2 weeks (14±7 days) after end of build-up period for each patient under both treatments within two time periods with each a length of 4 weeks
Pharmacogenetic analysis | 4 weeks
  Number of patients with SNPs in selected genes (CYP3A4, CYP3A5, ABCD1)
Tacrolimus trough levels | 4 weeks
  Tacrolimus trough levels in ng/mL, compared intra- and interindividually.
Doses of prolonged-release tacrolimus | 4 weeks
  Doses of prolonged-release tacrolimus (Envarsus®) in ng/mL.
Number of patients with adverse event or toxicity | 10 weeks
  Cumulative dosage and signs of tacrolimus toxicity and adverse events. Potentially tacrolimus associated adverse events and toxicity are recorded individually and compared with individual tacrolimus AUCs. Special attention is taken e.g. towards metabolic (elevated concentration of blood glucose, fat), hematopoetic (cell counts), neurological (tremor, headache), renal (change in glomerular filtration rate), gastrointestinal (diarrhea, nausea), hepatic (cholestasis, elevated transaminases, blood clotting disorder), elevated blood pressure.
Number of adverse events or toxicity per patient | 10 weeks
  Special attention is taken e.g. towards metabolic (elevated concentration of blood glucose, fat), hematopoetic (cell counts), neurological (tremor, headache), renal (change in glomerular filtration rate), gastrointestinal (diarrhea, nausea), hepatic (cholestasis, elevated transaminases, blood clotting disorder), elevated blood pressure.
eGFR (CKiD formula) | 4 weeks
  eGFR (CKiD formula) comparing the two study phases
Treatment failure rate | 10 weeks
  composite endpoint: any patient who experienced death, graft failure, BPAR or lost to follow-up
limited sampling strategy (LSS) | 4 weeks
  LSS driven 24h-AUC estimation
Taxonomy of the gut microbiome | 10 weeks
  Taxonomy of the gut microbiome using metagenomic sequencing
Gut microbial metabolism | 10 weeks
  Functional assessment of the gut microbiome using LC-MS based metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Lars Pape, Prof. Dr., Principal Investigator — University Hospital of Essen, Pediatrics II
Locations (4):
- Germany (4):
  - University Hospital Cologne, Pediatrics, Cologne
  - University Hospital of Essen, Pediatrics II, Essen
  - University Hospital of Hamburg-Eppendorf, Hamburg
  - University Hospital of Heidelberg, Heidelberg

REFERENCES:
- [Derived] Karaterzi S, Tonshoff B, Ahlenstiel-Grunow T, Baghai M, Beck B, Buscher A, Eifler L, Giese T, Lezius S, Muller C, Oh J, Zapf A, Weber LT, Pape L. A multi-center interventional study to assess pharmacokinetics, effectiveness, and tolerability of prolonged-release tacrolimus after pediatric kidney transplantation: study protocol for a prospective, open-label, randomized, two-phase, two-sequence, single dose, crossover, phase III b trial. Front Nephrol. 2024 Feb 20;4:1331510. doi: 10.3389/fneph.2024.1331510. eCollection 2024. PMID 38444519